CLINICAL TRIAL: NCT02644941
Title: An Assessment of Humacyte's Human Acellular Vessel in Patients Needing Renal Replacement Therapy: A Comparison With ePTFE Grafts as Conduits for Hemodialysis (HUMANITY)
Brief Title: Comparison of the Human Acellular Vessel (HAV) With ePTFE Grafts as Conduits for Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Humacyte, Inc. (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN-PRO-V006; 2015-003261-28 (EudraCT Number)
Record Dates: First submitted 2015-12-29; First posted 2016-01-01 (Estimated); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Renal Failure; End Stage Renal Disease; Hemodialysis; Vascular Access
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic | interventions — Social Control, Formal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human Acellular Vessel (HAV) (Experimental): HAV-tissue-engineered vascular conduit (6mm diameter)
  Interventions: Biological: Human Acellular Vessel (HAV)
- ePTFE (Active Comparator): One of two commercially available comparators (Bard Impra® and Gore PROPATEN®)
  Interventions: Device: ePTFE graft

INTERVENTIONS:
Biological: Human Acellular Vessel (HAV) — HAV-tissue-engineered vascular conduit (6mm diameter)
  Other Names: (regulated as a biological product)
  Arms: Human Acellular Vessel (HAV)
Device: ePTFE graft — One of two commercially available comparators (Bard Impra® and Gore PROPATEN®)
  Arms: ePTFE

SUMMARY:
The main purpose of this study is to compare the Human Acellular Vessel (HAV) with ePTFE grafts when used for hemodialysis access.

DETAILED DESCRIPTION:
This is a Phase 3, prospective, multicenter, multinational, open-label, randomized, two-arm, comparative study. Subjects who sign informed consent would undergo study-specific screening assessments within 35 days from the day of informed consent.

Participants who consented were randomized to the HAV treatment arm of one of the two commercially available comparators.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ESRD who need placement of an AV graft in the arm.
* Either on hemodialysis or expected to start hemodialysis within 12 weeks of study conduit implantation.
* Suitable anatomy for implantation of straight or looped conduits in either the forearm or upper arm (not crossing the elbow).
* Hemoglobin ≥8 g/dL and platelet count ≥100,000 cells/mm3 prior to Day 0 (within 35 days).
* Other hematological and biochemical parameters within a range consistent with ESRD prior to Day 0 (within 35 days).
* Adequate liver function prior to Day 0 (within 35 days).
* Female subjects must be either:

  * Of non-childbearing potential Or
  * Must agree to use at least one form of birth control methods for the duration of the study.
* Subject, or legal representative, able to communicate effectively with investigative staff, competent and willing to give written informed consent, and able to comply with entire study procedures including all scheduled follow-up visits.
* Life expectancy of at least 1 year.

Exclusion Criteria:

* History or evidence of severe peripheral vascular disease in the intended arm for implantation.
* Known or suspected central vein stenosis or conduit occlusion on the ipsilateral side of planned implantation, unless the stenosis is corrected prior to study conduit implantation.
* Treatment with any investigational drug or device within 60 days prior to study entry (Day 0).
* Cancer that is actively being treated with a cytotoxic agent.
* Documented hyper-coagulable state.
* Bleeding diathesis.
* Active clinically significant immune-mediated disease, not controlled by maintenance immunosuppression.
* High dose glucocorticoid therapy for treatment of autoimmune flare, or other inflammatory diseases is excluded.
* Patients using glucocorticoids for immunosuppression post-transplant to prevent against transplanted allograft rejection in the period post allograft failure are excluded.
* The following examples of immunosuppressive agents (or the like) are exclusionary for enrollment in this clinical trial:
* tacrolimus or FK506 [Prograf]
* mycophenolate mofetil [Cellcept],
* cyclosporine [Sandimmune or Gengraf] i-Sirolimus administered systemically (Sirolimus in drug eluting stents is NOT an exclusion)
* Anticipated renal transplant within 6 months.
* Venous outflow from study conduit cannot be placed more centrally than the venous outflow of any previous failed access in that extremity.
* Active local or systemic infection (white blood cells [WBC] > 15,000 cells/mm3 at Screening). If the infection resolves, the subject must be at least one week post resolution of that infection before implantation.
* Known serious allergy to planned antiplatelet agent.
* Pregnant women, or women intending to become pregnant during the course of the trial.
* Any other condition which in the judgment of the investigator would preclude adequate evaluation of the safety and efficacy of the study conduit.
* Previous enrollment in this study or any other study with the HAV.
* Employees of Humacyte and employees or relatives of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2023-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shamik Parikh, MD, Study Director — Humacyte, Inc.
Locations (38):
- United States (22):
  - Arizona Kidney Disease and Hypertension Center (AKDHC), Phoenix, Arizona
  - Carondelet St. Mary's Hospital, Tucson, Arizona
  - Ladenheim Dialysis Access Center, Fresno, California
  - General Surgery and Vascular Access, Fresno, California
  - University of California Irvine (UCI) Medical Center, Irvine, California
  - VA Long Beach Healthcare System, Long Beach, California
  - VA Sacramento Medical Center, Mather, California
  - Balboa Nephrology, San Diego, California
  - University of South Florida, Tampa, Florida
  - Southwest Vascular Access Center, Alsip, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Cardiovascular Institute, Flint, Michigan
  - Greenwood Leflore Hospital, Greenwood, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers-New Jersey Medical School, Newark, New Jersey
  - The Cardiovascular Care Group, Westfield, New Jersey
  - Duke University Hospital, Durham, North Carolina
  - Kaiser Permanente, Portland, Oregon
  - Medical University of South Carolina (MUSC), Orangeburg, South Carolina
  - Baylor Scott and White Research Institute, Dallas, Texas
  - University of Wisconsin, Madison, Wisconsin
- Germany (2):
  - Universitätsklinikmn Erlangen, Gefäßchirurgie - Chirurgisches Zentrum, Erlangen, Bavaria
  - Universitätsklinikum Frankfurt Klinik für Gefäß- und Endovascular-Chirurgie, Frankfurt am Main, Hesse
- Israel (5):
  - The Chaim Sheba Medical Center, Ramat Gan, Tel Aviv
  - Hillel Jaffe Medical Center, Hadera
  - Rambam Health Care Campus, Haifa
  - Sharee Zedek Medical Center, Jerusalem
  - Yitzhak Shamir Medical Center - Assaf Harofeh, Tzrifin
- Poland (3):
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego, Poznan
  - Samodzielny Publiczyn Centralny Szpital Klinziczny w Warszawie - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego, Warsaw
  - Wojewódzki Szpital Specjalistyczny we Wrocławiu, Wroclaw
- Grupo de Estudos Vasculares, Porto, Portugal
- United Kingdom (5):
  - Leicester General Hospital, Leicester, East Midlands/ Leicestershire
  - Guy´s Hospital, Kings´College London, London, Greater London
  - Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands
  - Queen Elizabeth University Hospital Glasgow, Glasgow
  - Leeds General Infirmary, Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Blalock SKF, Levitan GS, Prichard HL, Niklason LE, Kirkton RD. Biological mechanisms of infection resistance in tissue engineered blood vessels compared to synthetic expanded polytetrafluoroethylene grafts. JVS Vasc Sci. 2023 Jul 14;4:100120. doi: 10.1016/j.jvssci.2023.100120. eCollection 2023. PMID 37662589

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a large multicenter comparative study conducted at 37 centers in 6 countries to compare the HAV and ePTFE.
Groups:
- ePTFE: The comparator is one two commercially available 6 mm ePTFE grafts (Bard Impra® or Gore PROPATEN®)
Period: 18 Months
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Started | 177 | 178
Completed | 128 | 126
Not Completed | 49 | 52
Not completed — Subjects lost graft during the study up to the data cut-off | 49 | 52
Period: 24 Months
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Started | 177 | 178
Completed | 108 | 106
Not Completed | 69 | 72
Period: 60 Months
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Started | 177 | 178
Completed | 78 | 80
Not Completed | 99 | 98

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Human Acellular Vessel (HAV) | ePTFE | Total
Number analyzed (Participants) | 177 | 178 | 355
Age, Customized [Number; unit: Age range of participants]
  18-21 years | 0 | 1 | 1
  22-44 years | 21 | 22 | 43
  45-64 years | 69 | 78 | 147
  65-74 years | 57 | 50 | 107
  >/= 75 years | 30 | 27 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 90 | 179
  Male | 88 | 88 | 176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 20 | 46
  Not Hispanic or Latino | 129 | 127 | 256
  Unknown or Not Reported | 22 | 31 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 123 | 116 | 239
  Black or African American | 44 | 49 | 93
  Asian | 4 | 6 | 10
  American Indian or Alaska Native | 4 | 3 | 7
  Other | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 103 | 103 | 206
  Europe | 62 | 61 | 123
  Israel | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Loss of Secondary Patency
Description: 1. Defined as 'the interval from the time of access placement until access abandonment', i.e., patent with or without interventions (Sidawy et al. 2002).
  2. "Abandonment" defined as no remaining segment of the study conduit was incorporated into the vascular access circuit used for dialysis (conversely, if some portion of the study conduit was still being used for dialysis it was not considered abandoned).
Time Frame: 12 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 29 | 34

2. Primary Outcome: Number of Participants With Loss of Secondary Patency
Description: as for outcome 1
Time Frame: 18 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 41 | 37

3. Primary Outcome: Number of Participants With Loss of Secondary Patency
Description: as for outcome 1
Time Frame: 24 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 48 | 41

4. Secondary Outcome: Number of Participants With Loss of Primary Patency
Description: Use of duplex ultrasonography to assess study conduit patency. Loss of primary patency occurs when any intervention is performed on the conduit regardless of whether the conduit thrombosed.
Time Frame: 12 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 118 | 78

5. Secondary Outcome: Number of Participants With Loss of Primary Patency
Description: as for outcome 4
Time Frame: 18 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 146 | 111

6. Secondary Outcome: Number of Participants With Loss of Primary Patency
Description: as for outcome 4
Time Frame: 24 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 132 | 104

7. Secondary Outcome: Number of Participants With Loss of Primary Patency
Description: Duplex ultrasound was used to assess study conduit patency. Loss of primary patency occurs when any intervention is performed on the conduit regardless of whether the conduit thrombosed.
Time Frame: 60 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 146 | 121

8. Secondary Outcome: Study Conduit Abandonment
Description: No remaining segment of the study conduit is incorporated into the vascular access circuit used for dialysis.
Time Frame: 24 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 57 | 44

9. Secondary Outcome: Study Conduit Abandonment
Description: No remaining segment of the study conduit is incorporated into the vascular access circuit used for dialysis.
Time Frame: 60 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 69 | 53

10. Secondary Outcome: Rate of Adjudicated Study Conduit Access Related Infections
Description: Adjudicated using the standard definition of access-related infections (CDC; 2013).
Time Frame: 24 months post-implantation
Measure: Number; unit: Events per 100 Person-Years
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Events per 100 Person-Years | 0.93 | 4.54

11. Secondary Outcome: Access-related Infections
Description: Using Dialysis Event Surveillance Manual: CDC; 2013.
Time Frame: 60 months post-implantation
Measure: Number; unit: Access related infection events
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Access related infection events | 17 | 27

12. Secondary Outcome: Participants With at Least 1 Intervention Required to Achieve/Maintain Secondary Patency
Description: Rate of intervention defined as the number of interventions per participant per year while conduit is patent (i.e., has not been abandoned).
  Number of successful interventions to achieve/maintain Secondary Patency.
Time Frame: 24 months post-implantation
Measure: Count of Participants; unit: Participants
Groups:
- ePTFE: One of two commercially available comparator (Bard Impra® and Gore PROPATEN®)
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 146 | 116

13. Secondary Outcome: Total Interventions Performed to Maintain Secondary Patency (Ballon Size Not > 6 Millimeters)
Description: Total number of interventions performed by treatment group stratified by any use of balloon size no > 6 millimeters.
Time Frame: 60 months post-implantation
Population: Non-oversized ballon use (no greater than 6 mm)
Measure: Mean (Standard Deviation); unit: Interventions per participant
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Interventions per participant | 2.7 (3.68) | 2.7 (3.77)

14. Secondary Outcome: Total Interventions Performed to Maintain Secondary Patency (Balloon Size > 6 Millimeters)
Description: Total number of interventions performed by treatment group stratified by any use of balloon size greater than 6 millimeters.
Time Frame: 60 months post-implantation
Population: Oversized ballon use (greater than 6 mm)
Measure: Mean (Standard Deviation); unit: Interventions per participant
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Interventions per participant | 7.3 (5.74) | 2.7 (3.77)

15. Secondary Outcome: Thrombosis of Study Access That Required Intervention
Description: Total number of thrombosis events (per each treatment group) that required an intervention to maintain the functionality of patent access
Time Frame: 24 months post-implantation
Measure: Number; unit: Thrombosis events requiring intervention
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Thrombosis events requiring intervention | 361 | 170

16. Secondary Outcome: Thrombosis of Study Access That Required Intervention
Description: as for outcome 15
Time Frame: 60 months post-implantation
Measure: Number; unit: Thrombosis events requiring intervention
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Thrombosis events requiring intervention | 409 | 205

17. Secondary Outcome: Dialysis Efficiency as Measured by spKt/Vurea (Subset of Subjects)
Description: Dialysis efficiency as assessed by spKt/Vurea (obtained from dialysis unit for a subset of subjects) will be summarized descriptively. The most recent available data prior to the study visits will be used for the analysis.
  Twenty sites provided at least 1 spKt/Vurea measurement. spKt/Vurea: measure of dialysis adequacy for a single hemodialysis treatment using the single pooled method.
Time Frame: 2 to 18 Months post-implantation
Population: Female and Male
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 69 | 72
unitless | 1.61 (0.551) | 1.67 (0.445)

18. Secondary Outcome: Severity of Adverse Events
Description: Severity Assessment Standard
  1. Mild: Events require minimal or no treatment and do not interfere with the subject's daily activities.
  2. Moderate: Events result in a low level of inconvenience or concern with the therapeutic measures. May cause some interference with functioning.
  3. Severe: Events interrupt a subject's usual daily activity and may require systemic drug therapy or other treatment. Severe events are usually incapacitating.
  4. Life-threatening: Any adverse event that places the subject or participant, in the view of the investigator, at immediate risk of death from the reaction as it occurred, i.e., it does not include a reaction that, had it occurred in a more severe form, might have caused death.
  5. Death: Death related to Adverse Event.
Time Frame: 24 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants
  Mild | 8 | 9
  Moderate | 39 | 55
  Severe | 74 | 64
  Life-threatening | 9 | 7
  Death | 45 | 39

19. Secondary Outcome: Number of Participants With at Least One Adverse Event
Description: Collection of all Adverse Events beginning on Day 0 after implantation up to 2 years post implantation (Month 24).
Time Frame: 24 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 175 | 174

20. Secondary Outcome: True Aneurysm Formation (Conduit Lumen Diameter >9 Millimeters)
Description: Assessed by ultrasound: at least a 50% increase over the 6 millimeter baseline
Time Frame: 24 months post-implantation
Measure: Number; unit: Total number of aneurysms
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Total number of aneurysms | 19 | 11

21. Secondary Outcome: True Aneurysm Formation (Conduit Lumen Diameter >9 Millimeters)
Description: Assessed by ultrasound: at least a 50% increase over the 6 millimeter baseline
Time Frame: 60 months post-implantation
Measure: Number; unit: Total number of aneurysms
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Total number of aneurysms | 23 | 12

22. Secondary Outcome: Pseudoaneurysm Formation
Description: Use of duplex ultrasound to assess the diameter of the lumen mid-conduit. The outcome measures data represents the total number of pseudoaneurysms.
Time Frame: 24 months post-implantation
Measure: Number; unit: Pseudoaneurysms
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Pseudoaneurysms | 98 | 47

23. Secondary Outcome: Pseudoaneurysm Formation
Description: as for outcome 22
Time Frame: 60 months post-implantation
Measure: Number; unit: Pseudoaneurysms
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Pseudoaneurysms | 113 | 59

24. Secondary Outcome: Study Conduit Spontaneous Ruptures Due to Iatrogenic Injury
Description: Assessed by ultrasound
Time Frame: 24 months post-implantation
Measure: Number; unit: Ruptures d/t iatrogenic injury
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Ruptures d/t iatrogenic injury | 0 | 0

25. Secondary Outcome: Study Conduit Spontaneous Ruptures Due to Iatrogenic Injury
Description: Assessed by ultrasound
Time Frame: 60 months post-implantation
Measure: Number; unit: Ruptures d/t iatrogenic injury
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Ruptures d/t iatrogenic injury | 0 | 0

26. Secondary Outcome: Anastomotic Bleeding or Rupture
Description: Assessed by ultrasound
Time Frame: 24 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 0 | 0

27. Secondary Outcome: Anastomotic Bleeding or Rupture
Description: Assessed by ultrasound
Time Frame: 60 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 0 | 0

28. Secondary Outcome: Calculated Panel Reactive Antibody More Than 20% Change From Baseline
Description: Increase in Panel Reactive Antibody more than 20% (highly sensitized) from baseline
Time Frame: 18 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 3 | 8

29. Secondary Outcome: Calculated Panel Reactive Antibody More Than 20% Change From Baseline
Description: Increase in Panel Reactive Antibody more than 20% (highly sensitized) from baseline
Time Frame: 24 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Participants | 2 | 10

30. Secondary Outcome: Mean Inner Diameter of Conduit (Millimeter)
Description: Duplex ultrasonography: diameter of the mid-conduit lumen
Time Frame: 12 months post-implantation
Measure: Mean (Standard Deviation); unit: Inner diameter (millimeter)
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Inner diameter (millimeter) | 6.20 (1.452) | 5.66 (1.601)

31. Secondary Outcome: Mean Inner Diameter of Conduit (Millimeter)
Description: Duplex ultrasonography: diameter of the mid-conduit lumen
Time Frame: 24 months post-implantation
Measure: Mean (Standard Deviation); unit: Inner diameter (millimeter)
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Inner diameter (millimeter) | 6.02 (2.898) | 5.88 (2.209)

32. Secondary Outcome: Mean Inner Diameter of Conduit (Millimeter)
Description: Duplex ultrasonography: diameter of the mid-conduit lumen
Time Frame: 60 months post-implantation
Measure: Mean (Standard Deviation); unit: Inner diameter (millimeter)
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
Number analyzed (Participants) | 177 | 178
Inner diameter (millimeter) | 6.19 (1.979) | 6.23 (1.131)

ADVERSE EVENTS:
Time Frame: All study participants were followed to 24 months post-implantation at routine study visits regardless of patency status. After 24 months, participants with a patent study conduit were followed (while the study conduit remained patent) for up to 5 years (60 months) post-implantation at routine study visits.
Arm/Group | Human Acellular Vessel (HAV) | ePTFE
All-Cause Mortality (participants affected / at risk) | 46/177 | 39/178
Serious Adverse Events (participants affected / at risk) | 157/177 | 146/178
Other Adverse Events (participants affected / at risk) | 176/177 | 176/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Acellular Vessel (HAV) (N=177) | ePTFE (N=178)
Anemia (Blood and lymphatic system disorders) | 7 (9) | 10 (13)
Cardiac arrest (Cardiac disorders) | 6 (38) | 11 (32)
Cardiac failure congestive (Cardiac disorders) | 6 (38) | 8 (32)
Pneumonia (Infections and infestations) | 11 (61) | 18 (72)
Sepsis (Infections and infestations) | 13 (61) | 12 (72)
Vascular access site infection (Infections and infestations) | 13 (61) | 18 (72)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 17 (99) | 5 (71)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 81 (99) | 57 (71)
Hyperkalemia (Metabolism and nutrition disorders) | 9 (21) | 9 (26)
Hypotension (Vascular disorders) | 10 (77) | 4 (69)
Vascular stenosis (Vascular disorders) | 53 (77) | 49 (69)
Venous stenosis (Vascular disorders) | 7 (78) | 9 (74)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Acellular Vessel (HAV) (N=177) | ePTFE (N=178)
Anemia (Blood and lymphatic system disorders) | 19 (31) | 19 (30)
Abdominal pain (Gastrointestinal disorders) | 8 (51) | 10 (53)
Diarrhea (Gastrointestinal disorders) | 15 (51) | 10 (53)
Nausea (Gastrointestinal disorders) | 12 (51) | 17 (53)
Vomiting (Gastrointestinal disorders) | 13 (51) | 12 (53)
Edema peripheral (General disorders) | 9 (72) | 14 (81)
Implant site extravasation (General disorders) | 11 (72) | 11 (81)
Peripheral swelling (General disorders) | 13 (72) | 8 (81)
Pneumonia (Infections and infestations) | 18 (90) | 23 (105)
Sepsis (Infections and infestations) | 14 (90) | 12 (105)
Upper respiratory infection (Infections and infestations) | 8 (90) | 11 (105)
Urinary tract infection (Infections and infestations) | 16 (90) | 12 (105)
Vascular access site infection (Infections and infestations) | 17 (90) | 27 (105)
Vascular access site hematoma (Injury, poisoning and procedural complications) | 48 (168) | 37 (150)
Vascular access site hemorrhage (Injury, poisoning and procedural complications) | 43 (168) | 35 (150)
Vascular access edema (Injury, poisoning and procedural complications) | 9 (168) | 9 (150)
Vascular access site pain (Injury, poisoning and procedural complications) | 13 (168) | 18 (150)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 75 (168) | 41 (150)
Vascular access site swelling (Injury, poisoning and procedural complications) | 28 (168) | 21 (150)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 124 (168) | 93 (150)
Fluid overload (Metabolism and nutrition disorders) | 12 (55) | 11 (61)
Hyperkalemia (Metabolism and nutrition disorders) | 25 (55) | 26 (61)
Hypoglycemia (Metabolism and nutrition disorders) | 6 (55) | 12 (61)
Hypoesthesia (Nervous system disorders) | 8 (49) | 14 (56)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (54) | 10 (38)
Aneurysm (Vascular disorders) | 19 (156) | 12 (144)
Hypertension (Vascular disorders) | 9 (156) | 14 (144)
Hypotension (Vascular disorders) | 23 (156) | 12 (144)
Steal syndrome (Vascular disorders) | 19 (156) | 15 (144)
Subclavian vein stenosis (Vascular disorders) | 9 (156) | 9 (144)
Vascular stenosis (Vascular disorders) | 139 (156) | 123 (144)
Venous stenosis (Vascular disorders) | 24 (156) | 28 (144)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT02644941/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT02644941/SAP_001.pdf